CLINICAL TRIAL: NCT07207525
Title: Sources of Information and Search Patterns on Pulmonary Hypertension in Patients With Confirmed Diagnosis and Their Caregivers (inPHorma)
Brief Title: Information Sources in Pulmonary Hypertension
Acronym: inPHorma
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, PhD, University of Sao Paulo General Hospital
Other Study IDs: SGP 27368
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Pulmonary Hypertension; Patients; Information Needs; Information Sources; Health Information Seeking
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Pulmonary Hypertension: Adults (≥18 years) with a confirmed diagnosis of pulmonary hypertension, from any clinical group. Participants will complete a structured, self-administered questionnaire about their sources of health information, expectations, satisfaction, and preferred communication channels. No intervention or treatment is provided.
- Informal Caregivers of Pulmonary Hypertension Patients: Adults (≥18 years) who provide non-professional care or support to a patient with pulmonary hypertension (family member or close contact). Caregivers will complete the same structured questionnaire, focusing on their experiences, information needs, and trusted sources. No intervention or treatment is provided.

SUMMARY:
Pulmonary hypertension is a serious disease that affects patients' health, daily life, and emotional well-being. Many patients and their caregivers actively look for information to better understand the condition and its treatment. However, the quality of information found in different sources, such as the internet, social media, health professionals, and patient groups, can vary.

This study will use a short questionnaire to learn where patients and caregivers search for information, what topics they look for, how satisfied they are with what they find, and which sources they trust most. The results will help improve communication strategies, educational materials, and support programs for people living with pulmonary hypertension and their families.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a chronic and progressive disease often diagnosed late, which forces patients and caregivers to actively seek information to understand and manage the condition. The complexity of PH, combined with its physical, emotional, and social impact, makes access to reliable health information essential.

This cross-sectional observational study will apply a structured, self-administered questionnaire to approximately 200 participants (100 patients with confirmed PH and 100 informal caregivers). The questionnaire covers demographic and clinical characteristics, information sources used, expectations and satisfaction, most frequently searched topics, experiences with conflicting information, and preferred communication channels.

The goal is to describe patterns of health information seeking in this population and identify opportunities to improve communication, educational resources, and patient-caregiver support. Findings are expected to contribute to the development of more effective health communication strategies and to guide health professionals in addressing information needs in pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of pulmonary hypertension (any clinical group) or informal caregiver of a patient with pulmonary hypertension
* Ability to read and understand the questionnaire
* Signed informed consent (ICF/TCLE)

Exclusion Criteria:

* Inability to understand or complete the questionnaire
* Refusal to participate or not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a confirmed diagnosis of pulmonary hypertension and their informal caregivers (family members or non-professional supporters), recruited from a specialized center in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Main Sources of Health Information | Up to 12 months after study start
  Identification of the primary sources of information used by patients with pulmonary hypertension and their informal caregivers, as reported in the structured questionnaire.

SECONDARY OUTCOMES:
Satisfaction With Health Information | Up to 12 months after study start
  Level of satisfaction with the health information found, measured on a 5-point Likert scale (1 = not satisfied, 5 = very satisfied).
Confidence in Finding Information | Up to 12 months after study start
  Degree of confidence when searching for information, measured on a 5-point Likert scale (1 = not confident, 5 = very confident).
Frequency of Conflicting Information | Up to 12 months after study start
  Proportion of participants reporting that they found contradictory or inconsistent health information related to pulmonary hypertension.
Most Frequently Searched Topics | Up to 12 months after study start
  Distribution of the main topics searched (e.g., treatments, prognosis, daily care, rights/benefits) as reported in the questionnaire.
Trusted Communication Channels | Up to 12 months after study start
  Identification of the channels considered most reliable for health information (e.g., physician, healthcare team, patient groups, internet sources).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração (InCor), Hospital das Clínicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided